CLINICAL TRIAL: NCT01101334
Title: Phase 2 Study of CS-7017 and Erlotinib in Subjects With Advanced Non-Small Cell Lung Cancer Who Failed First Line Therapy
Brief Title: Study of Erlotinib With or Without Investigational Drug (CS-7017) in Subjects With Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS7017-A-U204
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Advanced Non-small Cell Lung Cancer (NSCLC)
Keywords: NSCLC
MeSH Terms: interventions — efatutazone; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CS-7017 plus erlotinib (Experimental)
  Interventions: Drug: CS-7017; Drug: erlotinib
- erlotinib (Active Comparator)
  Interventions: Drug: erlotinib

INTERVENTIONS:
Drug: CS-7017 — CS-7017, Two 0.25mg Tablets administered twice daily
  Arms: CS-7017 plus erlotinib
Drug: erlotinib — Erlotinib; One 150mg tablet administered once daily
  Other Names: Tarceva

SUMMARY:
This is a Phase 2 and open-label (subject will know the treatment he or she is receiving) study. The subject will receive either Erlotinib alone or Erlotinib + CS-7017 in this study.

The study will determine what effect adding CS-7017 to Erlotinib has on safety and length of survival in subjects with advanced non-small cell lung cancer who failed the first treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIB or IV NSCLC.
* Recurrent disease (either no response to treatment or subsequent relapse after an objective response) that has progressed after first line therapy.
* Measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 criteria.
* ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Adequate organ and bone marrow function.
* Resolution of any toxic effects of prior therapy (except alopecia) to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.0 grade ≤ 1.
* Agreement to use effective contraception while on treatment and for at least 3 months after end of treatment.

Exclusion Criteria:

* Treatment with anticancer therapy within 3 weeks before study treatment.
* Therapeutic or palliative radiation therapy within 2 weeks or major surgery within 4 weeks before study treatment (except for radiotherapy for brain metastases).
* Administration of other thiazolidinediones (TZDs) within 4 weeks before study treatment.
* Current need for concomitant use of other TZDs during the study.
* Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals, known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection at time of screening.
* History of any of the following conditions within 6 months before initiating study treatment: diabetes mellitus requiring treatment with insulin or TZD agents; myocardial infarction with significant impairment of cardiac function; severe/unstable angina pectoris; coronary/peripheral artery bypass graft; New York Heart Association (NYHA) class III or IV congestive heart failure; malabsorption syndrome, chronic diarrhea (lasting > 4 weeks), inflammatory bowel disease, or partial bowel obstruction.
* Pericardial or pleural effusion (eg, requiring drainage) or pericardial involvement with the tumor. Participants with minimal pleural effusion may be eligible upon request by Investigator and approval by Sponsor.
* Pregnant or breast feeding.
* Prior treatment with epidermal growth factor receptor (EGFR) inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (17):
- United States (3):
  - DHHA, Denver, Colorado
  - Gabrail Cancer Center, Canton, Ohio
  - Providence Regional Medical Center Everett, Everett, Washington
- Zentrum fur Pneumologie und Thoraxchirurgie, Gauting, Germany
- India (8):
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Vedanta Institute of Medical Sciences, Ahmedabad, Gujarat
  - Kodlikeri Memorial Hospital, Aurangabad, Maharashtra
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Noble Hospital, Pune, Maharashtra
  - Apollo Speciality Hospital, Chennai, Tamil Nadu
  - Meenakshi Mission Hospital, Madurai, Tamil Nadu
  - Orchid Nursing Home, Kolkata, West Bengal
- South Korea (5):
  - St. Vincent's Hospital, Gyeonggi-do
  - Hwasun Hospital, Jeonnam
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 90 participants who met all inclusion and no exclusion criteria were randomized to treatment; 89 participants received treatment.
Groups:
- CS-7017 Plus Erlotinib: Participants who received two 0.25 mg CS-7017 tablets administered twice daily and one 150 mg erlotinib tablet administered once daily.
- Erlotinib: Participants who received one 150 mg erlotinib tablet administered once daily.
Period: Overall Study
Arm/Group | CS-7017 Plus Erlotinib | Erlotinib
Started | 45 | 45
Received Study Treatment | 44 | 45
Completed | 0 | 0
Not Completed | 45 | 45
Not completed — Adverse Event | 9 | 4
Not completed — Death | 7 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Withdrawal by Sponsor | 1 | 1
Not completed — Progressive Disease | 22 | 35
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for all participants who received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | CS-7017 Plus Erlotinib | Erlotinib | Total
Number analyzed (Participants) | 44 | 45 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 31 | 64
  >=65 years | 11 | 14 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (10.36) | 61.4 (11.34) | 60.5 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 20 | 31
  Male | 33 | 25 | 58

OUTCOME MEASURES:

1. Primary Outcome: Summary of Analysis of Progression-Free Survival Following Administration of CS-7017 and Erlotinib in Participants With Advanced Non-Small Cell Lung Cancer Who Failed First Line Therapy
Description: Progression-free survival (PFS) was defined as the time from randomization date of the first objective documentation of disease progression or death resulting from any cause, whichever comes first.
Time Frame: Baseline to disease progression or death, up to approximately 2.5 years
Population: PFS was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CS-7017 Plus Erlotinib | Erlotinib
Number analyzed (Participants) | 44 | 45
months | 4.1 [2.7 to 6.7] | 3.0 [2.2 to 5.3]

2. Secondary Outcome: Analysis of Overall Survival Following Administration of CS-7017 and Erlotinib in Participants With Advanced Non-Small Cell Lung Cancer Who Failed First Line Therapy
Description: Overall survival (OS) was defined as the time from randomization until death from any cause.
Time Frame: Baseline to death, up to approximately 2.5 years
Population: OS was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CS-7017 Plus Erlotinib | Erlotinib
Number analyzed (Participants) | 44 | 45
months | 7.6 [3.8 to 12.0] | 11.4 [9.7 to 15.0]

3. Secondary Outcome: Overall Response Rate Following Administration of CS-7017 and Erlotinib in Participants With Advanced Non-Small Cell Lung Cancer Who Failed First Line Therapy
Description: The overall response rate (ORR) was defined as the proportion of participants who achieved best overall response of complete response (CR) or partial response (PR); ORR = CR + PR. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions, CR was defined as the disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Time Frame: Baseline to disease progression or death, up to approximately 2.5 years
Population: ORR was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | CS-7017 Plus Erlotinib | Erlotinib
Number analyzed (Participants) | 44 | 45
Participants | 9 | 9

4. Secondary Outcome: Summary of Treatment-Emergent Adverse Events (TEAEs) Occurring in ≥10% of Participants Following Administration of CS-7017 and Erlotinib in Participants With Advanced Non-Small Cell Lung Cancer Who Failed First Line Therapy
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event that had an onset date on or after the first dose of CS-7017 or erlotinib up to and including 30 days after the last dose of any study drug, or worsened in severity after the first dose of CS-7017 or erlotinib relative to the pre-treatment state.
Time Frame: Baseline to 30 days after last dose, up to approximately 2.5 years
Population: TEAEs were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | CS-7017 Plus Erlotinib | Erlotinib
Number analyzed (Participants) | 44 | 45
Participants
  Any TEAE | 44 | 43
  Blood and Lymphatic System Disorders | 18 | 4
  Anaemia | 16 | 3
  Cardiac Disorders | 7 | 2
  Eye Disorders | 8 | 3
  Gastrointestinal Disorders | 27 | 25
  Constipation | 10 | 3
  Diarrhea | 18 | 19
  Nausea | 5 | 7
  Stomatitis | 6 | 6
  General Disorders & Administration Site Conditions | 41 | 19
  Asthenia | 9 | 8
  Disease progression | 8 | 5
  Face edema | 10 | 0
  Fatigue | 9 | 5
  Noncardiac chest pain | 5 | 2
  Edema peripheral | 17 | 1
  Pyrexia | 9 | 3
  Infections and Infestations | 13 | 16
  Investigations | 15 | 12
  Weight increased | 7 | 1
  Metabolism and Nutrition Disorders | 27 | 15
  Decreased appetite | 18 | 10
  Hypokalemia | 7 | 1
  Musculoskeletal and Connective Tissue Disorders | 15 | 10
  Pain in extremity | 7 | 0
  Nervous System Disorders | 15 | 6
  Dizziness | 5 | 2
  Headache | 5 | 1
  Psychiatric Disorders | 6 | 5
  Respiratory, Thoracic, and Mediastinal Disoders | 25 | 17
  Cough | 5 | 3
  Dyspnea | 9 | 7
  Pleural effusion | 10 | 0
  Skin and Subcutaneous Tissue Disorders | 33 | 30
  Alopecia | 5 | 0
  Dermatitis acneiform | 15 | 9
  Dry skin | 5 | 7
  Pruritus | 9 | 11
  Rash | 11 | 15
  Swelling face | 5 | 1
  Vascular Disorders | 1 | 5

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event (TEAE) data were collected from time of signing the informed consent form to the end of study assessment and follow-up period (30 days after last dose of study drug), up to approximately 2.5 years.
Description: A TEAE was defined as an adverse event that had an onset date on or after the first dose of CS-7017 or erlotinib up to and including 30 days after the last dose of any study drug, or worsened in severity after the first dose of CS-7017 or erlotinib relative to the pre-treatment state. All-cause mortality includes all deaths caused by TEAEs.
Arm/Group | CS-7017 Plus Erlotinib | Erlotinib
All-Cause Mortality (participants affected / at risk) | 15/44 | 7/45
Serious Adverse Events (participants affected / at risk) | 24/44 | 16/45
Other Adverse Events (participants affected / at risk) | 44/44 | 43/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CS-7017 Plus Erlotinib (N=44) | Erlotinib (N=45)
Anaemia (Blood and lymphatic system disorders) | 5 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 4
Hematochezia (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 2
Death (General disorders) | 4 | 1
Disease progression (General disorders) | 8 | 5
Multi-organ failure (General disorders) | 1 | 0
Edema peripheral (General disorders) | 2 | 0
Pain (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Femoral arterial stenosis (Vascular disorders) | 0 | 1
Macroangiopathy (Vascular disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Vascular stenosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CS-7017 Plus Erlotinib (N=44) | Erlotinib (N=45)
Anaemia (Blood and lymphatic system disorders) | 16 | 3
Death (General disorders) | 4 | 1
Disease progression (General disorders) | 8 | 5
Fatigue (General disorders) | 9 | 5
Neutrophil count decreased (Investigations) | 3 | 0
Any Blood and Lymphatic System Disorders (Blood and lymphatic system disorders) | 18 | 4
Any Cardiac Disorders (Cardiac disorders) | 7 | 2
Any General Disorders & Administration Site Conditions (General disorders) | 41 | 19
Any Investigations (Investigations) | 15 | 12
Any Neoplasms Benign, Malignant, and Unspecified (Including Cysts and Polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Any Respiratory, Thoracic, and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 25 | 17
Any Skin and Subcutaneous Tissue Conditions (Skin and subcutaneous tissue disorders) | 33 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No